CLINICAL TRIAL: NCT02132000
Title: Efficacy and Tolerability of Toremifene or Tamoxifen Therapy in Premenopausal Estrogen and Progesterone Receptor Positive Breast Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fengxi Su (Other)
Responsible Party: Sponsor-Investigator, Fengxi Su, Chief of Breast cancer center in Sun Yat-Sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCSCO002
Record Dates: First submitted 2014-04-30; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer Patients in Premenopausal; Estrogen and/or Progesterone Receptor Positive
MeSH Terms: interventions — Toremifene; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tamoxifen (Active Comparator): tamoxifen,20mg/day
  Interventions: Drug: toremifene or tamoxifen
- toremifene (Experimental): toremifene,60mg/day
  Interventions: Drug: toremifene or tamoxifen

INTERVENTIONS:
Drug: toremifene or tamoxifen

SUMMARY:
In premenopausal women, endocrine adjuvant therapy for breast cancer primarily consists of tamoxifen alone or with ovarian suppressive strategies. Toremifene is a chlorinated derivative of tamoxifen, but with a superior risk-benefit profile. In this trial, we sought to compare the efficacy and tolerability of toremifene and tamoxifen therapy in premenopausal patients with operable,estrogen and/or progesterone receptor positive breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Breast cancer
* Received standard treatment (chemotherapy, operation, or radiotherapy)
* premenopausal
* estrogen and/or progesterone receptor positive

Exclusion Criteria:

* Metastatic tumors
* During pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3036 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
survival outcomes: disease free survival | up to 5 years
5-year overall survival | up to 5 years

SECONDARY OUTCOMES:
side effects effects of therapies | Follow-up period,up to 5 years
  the primary safety measures are Hepatic function and blood lipid
Incidence of adverse events | follow-up period, up to 5 years
  Adverse events including hot flashes, irregular menses and others.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer center of Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China